CLINICAL TRIAL: NCT06629337
Title: Effect of Aerobic Exercise with Blood Flow Restriction on Post-exercise Hypotension in Young Adults: the Role of Histamine Receptors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Principal Investigator, Jong-Kyung Kim, Professor, California Baptist University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 141-2324-EXP
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Prehypertension (elevated Blood Pressure) or Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — fexofenadine; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: BFR exercise with histamine blockade (Experimental)
  Interventions: Genetic: H1 receptor blockade: 540 mg (Allegra), H2 receptor blockade: 40 mg (Pepcid AC)
- Sham Comparator: BFR exercise without histamine blockade (Sham Comparator)
  Interventions: Genetic: H1 receptor blockade: 540 mg (Allegra), H2 receptor blockade: 40 mg (Pepcid AC)

INTERVENTIONS:
Genetic: H1 receptor blockade: 540 mg (Allegra), H2 receptor blockade: 40 mg (Pepcid AC) — Subjects ingested fexofenadine (540 mg, tablet) at least 50 minutes before and famotidine (40 mg, tablet) 1 hour 50 minutes before the onset of each protocol because these dose of oral fexofenadine and famotidine reaches its peak concentration at around 1 h and 2 h, respectively

SUMMARY:
It was hypothesized that aerobic exercise with blood flow restriction (BFR) induced post exercise hypotension (PEH), and the reduction in blood pressure (BP) was due to peripheral vasodilation via the histamine receptors. Ten male participants participated in this study. The participants were randomly assigned to walk for 10 minutes at 6.4 k/m, 0% grade with or without BFR after taking histamine receptor blockade. Following exercise, BP was measured at 10 min interval for 60 minutes. Heart rate (HR), stroke volume (SV), cardiac output (CO), mean arterial pressure (MAP), and total peripheral resistance (TPR) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* good health,
* nonsmokers
* those not taking medications that could affect cardiovascular function

Exclusion Criteria:

* hypertension
* muscular skeletal disorder

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Post-exercise hypotension before and after the histamine blockade | 10 min, 20 min, 30 min, 40 min, 50 min, and 60 min post exercise
  Blood pressure change during 60 min (10 min interval) after BFR exercise

CONTACTS AND LOCATIONS:
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided